CLINICAL TRIAL: NCT03520985
Title: Alternate Day Dosing of Pomalidomide in Patients With Refractory Multiple Myeloma. A Multi-center, Single Arm Phase II Trial
Brief Title: Alternate Day Dosing of Pomalidomide in Patients With Refractory Multiple Myeloma
Acronym: OptiPOM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility (low patient accrual and financial reasons)
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 39/16 - OptiPOM
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Refractory Multiple Myeloma
Keywords: refractory Multiple Myeloma; Phase II; Pomalidomide; OptiPOM
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide (Experimental): The treatment in this trial consists of oral pomalidomide on alternate days (ad) plus Low-Dose Dexamethasone (adPOM + LD-DEX)
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide (4 mg p.o.) will be administered on every other day of each 28-day treatment cycle.
  Treatment duration:
  Treatment cycles are repeated until confirmed disease progression.
  Other Names: Imnovid®
Drug: Dexamethasone — For patients ≤ 75 years of age:
  Low-Dose Dexamethasone (40 mg p.o.) will be administered once per day on days 1, 7, 15, and 21 of a 28-day cycle.
  For patients > 75 years of age:
  Low-Dose Dexamethasone (20 mg p.o.) will be administered once per day on days 1, 7, 15, and 21 of a 28-day cycle.
  Treatment duration:
  Treatment cycles are repeated until confirmed disease progression.

SUMMARY:
Pomalidomide is an approved treatment for refractory multiple myeloma. Toxicity of pomalidomide in the pivotal MM-003 trial, was considerable, with 60% of patients experiencing drug-related G3/4 toxicity. Neutropenia (48% vs 16%) and pneumonia (13% vs 8%) were significantly more common in the pomalidomide arm. This resulted in frequent dose interruptions (67%) and dose reductions (27%). This suggests that for the majority of patients the 4 mg daily dosing schedule is too toxic, and that strategies to deliver reduced dosing of pomalidomide are of high practical relevance. The aim of this trial therefore is to establish that alternate day dosing of pomalidomide (4 mg q2d, d1-28) is non-inferior to daily dosing (4 mg d1-21 q28) in terms of efficacy of the drug with potentially less side effects.

DETAILED DESCRIPTION:
Multiple myeloma (MM) accounts for 1% of all cancers and ∼10% of all hematological malignancies. Despite recent advances in myeloma treatment, including the introduction of proteasome inhibitors, immunomodulatory drugs (IMiDs) and stem cell transplantation, myeloma remains an incurable disease. The treatment of bortezomib and lenalidomide refractory myeloma is still an unmet medical need. Once patients have relapsed after IMiD-containing therapies and have become bortezomib-resistant, their prognosis is extremely poor.

Pomalidomide is a third-generation, Swissmedic approved, oral immunomodulatory drug with activity in such patients. However the toxicity of pomalidomide in the pivotal MM-003 trial was considerable, with 60% of patients experiencing drug-related G3/4 toxicity. Neutropenia (48% vs 16%) and pneumonia (13% vs 8%) were significantly more common in the pomalidomide arm. This resulted in frequent dose interruptions (67%) and dose reductions (27%). This suggests that for the majority of patients the 4 mg daily dosing schedule (4 mg daily on 21 of 28 days) is toxic, and that strategies to deliver reduced dosing of pomalidomide are of high practical relevance.

Alternative dosing schedules:

There is robust data available indicating that lower pomalidomide doses (e.g. 2 mg daily) lead to similar responses and progression free survival with fewer side effects. Due to its unique pharmacological characteristics, pomalidomide is well suited for alternate day dosing. The decline of the plasma concentration at the terminal phase is slow. These data make pomalidomide an ideal candidate for alternate day dosing. Therefore, a phase I study has already been conducted in 2008 to test the alternating administration of the drug showing excellent responses with a marked reduction of thrombotic events and less severe myelosuppression.

The drug costs of pomalidomide are quite high. Interestingly, the manufacturer determined a pricing model that is independent from the capsule strength (costs for one capsule 1 mg=2 mg=3 mg=4 mg). In patients requiring dose reductions due to hematologic toxicity, daily dosing of reduced strength pomalidomide (e.g. 2 mg daily) is approved and suggested by the manufacturer. This delivers 50% less pomalidomide to the patient, albeit at 100% of the price of full dosing.

In summary, the establishment of the modified pomalidomide schedule would be an interesting option for our patients to achieve similar efficacy with fewer side effects. In addition, it would optimize the cost-effectiveness of the drug.

ELIGIBILITY:
Key inclusion criteria:

* Patient was diagnosed with multiple myeloma based on standard IMWG criteria
* Prior treatment with ≥ 2 treatment lines of anti-myeloma therapy
* Patients must have been exposed to both lenalidomide and bortezomib
* Measurable disease for myeloma defined as one of the following: serum M-protein ≥ 5 g/L; urine M-protein ≥ 0.2 g/24 hours
* Refractory or relapsed and refractory disease defined as documented disease progression during or within 60 days of completing their last myeloma therapy.
* Adequate hematological and hepatic function
* A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential

Key exclusion criteria:

* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration, with the exception of pT1-2 prostate cancer Gleason score ≤6, adequately treated, cervical carcinoma in situ or localized non-melanoma skin cancer.
* Polyneuropathy grade > 2
* Patients who received any of the following within the last 14 days of initiation of trial treatment:

  * Plasmapheresis
  * Major surgery (kyphoplasty is not considered major surgery)
  * Radiation therapy
  * Use of any anti-myeloma drug therapy
* Known or clinically suspected myeloma manifestations in the central nervous system
* Severe or uncontrolled cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of registration until 28 days after last dose of trial medication with longest treatment time of approximately 36 months
  OR is defined as minimal response or better, assessed according to the IMWG criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of registration until 28 days after last dose of trial medication with longest treatment time of approximately 36 months
  OS is defined as the time from registration until death from any cause. Patients not having an event at the time of analysis will be censored at the date they were last known to be alive.
Overall Survival (OS) at 12 months | at 12 months
  OS, as defined above, will be evaluated at 12 months.
Progression-free survival (PFS) | From date of registration until 28 days after last dose of trial medication with longest treatment time of approximately 36 months
  PFS is defined as the time from registration until progression according the IMWG criteria or death from any cause, whichever occurs first. Patients not having an event at the time of analysis as well as patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting a new treatment, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Zander, MD, Study Chair — Luzerner Kantonsspital; Christoph Driessen, Prof, Study Chair — Cantonal Hospital of St. Gallen; Christoph Renner, Prof, Study Chair — Onkozentrum Zürich
Locations (16):
- Switzerland (16):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden (Baden/Brugg), Baden
  - Universitätsspital Basel, Basel
  - Istituto Oncologico Svizzera Italiana IOSI, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hopital Fribourgeois HFR, Fribourg
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Luzerne
  - Spital Thurgau AG, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Regionalspital Thun, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum Hirslanden Zürich, Zurich
  - OnkoZentrum Zürich AG - Klinik im Park, Zurich
  - Universitätsspital Zürich, Zurich